CLINICAL TRIAL: NCT06253104
Title: Changes in Skeletal Muscle Thickness in Patients With Acute Heart Failure
Status: Recruiting | Type: Observational
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00004088
Record Dates: First submitted 2024-01-19; First posted 2024-02-12 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Heart Failure; Muscle Atrophy; Skeletal Muscle Atrophy; Cardiogenic Shock
MeSH Terms: conditions — Heart Failure; Muscular Atrophy; Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Study Cohort: All enrolled participants with no randomization group allocations
  Interventions: Diagnostic Test: BodyMetrix Body Composition Ultrasound

INTERVENTIONS:
Diagnostic Test: BodyMetrix Body Composition Ultrasound — We will use a BodyMetrix Pro A-mode ultrasound device (BodyMetrix Pro, Intelametrix Inc., Livermore, CA) which is a lay imaging tool designed specifically to assess body composition. Images will be taken at two sites; the lateral thigh and bicep on the dominant side if able to identify, or else on the right side. On each visit, five images will be taken at each site (the lateral thigh and bicep). Participants will be measured 2-3 days from initiation in study, then 7 days after, and then weekly from the first measurement until time of advanced therapy, discharge, or death. This measurement sequence will then be repeated following advanced therapy up until discharge or death. Each measurement session will last about 20-30 minutes. This will be performed by the PI or members of the study team who have been trained by the research coordinator.

SUMMARY:
This study aims to determine, via skeletal muscle ultrasound (US), the extent, timing and relationship between skeletal muscle mass loss and outcomes after orthotropic heart transplantation (OHT) and left ventricular assist device (LVAD) implantation amongst patients with cardiogenic shock. Advanced therapies such as OHT and VADs in the heart failure (HF) population may promote skeletal muscle mass and subsequent quality of life, but there is a lack of literature assessing muscle mass changes in HF patients before and after advanced therapies using US imaging. Therefore this observational study will provide further insight into the 1) changes in lean body mass during critical illness and 2) the feasibility of using bedside US to assess lean body mass in the inpatient setting.

DETAILED DESCRIPTION:
The investigators will be recruiting subjects with advanced cardiomyopathy in cardiogenic shock in the inpatient setting. This is an observational study to better understand changes in lean body mass during critical illness through a quick, safe, and non-invasive method. This study will also validate the use of the BodyMetrix BX 2000 Pro ultrasound machine for the assessment of body composition, particularly muscle wasting, in the cardiogenic shock population.

The ultrasound device received 501(k) designation from the FDA in 2009 for measurement of localized fat and muscle thickness. Baseline US muscle thickness assessments will occur at baseline after consent; then days 3 and 7 after baseline study visit; then every 7 days thereafter until end of the index hospitalization (discharge or death). Each measurement session will take about 20-30 minutes.The investigators will take measurements at two sites: the lateral thigh and bicep (participant's dominant side). Clear ultrasound gel will be applied to the skin and the ultrasound probe placed against the skin, and the muscle thickness measurement made five times at each position.

The US images are read after a study visit completion, with measurements taken at pre-specified anatomic landmarks to obtain the muscle thickness, which is averaged accross the duplicate measurements. The primary endpoints are: Percentage change in skeletal muscle thickness from admission to nadir; Percentage change in skeletal muscle thickness after advanced therapies; and the Relationship between muscle mass loss during cardiogenic shock and subsequent clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years of age
2. Ejection fraction <40%
3. Cardiogenic shock defined by clinical criteria (including any of: lactate >2.5 mmol/L, systolic blood pressure <90 mmHg, acute kidney or liver injury, or cardiac index <2.1 on hemodynamic monitoring) plus the clinical requirement for at least one pressor, inotrope, or temporary mechanical circulatory support device (MCSD)

Exclusion Criteria:

1. History of LVAD or other durable ventricular assist device
2. An identified clinical disorder associated with skeletal muscle weakness/wasting (e.g., muscular dystrophy, mitochondrial disorder, active cancer, modified Rankin score greater or equal to 4 post-stroke
3. Chronic enteric and parenteral nutrition support patients

Intubation or prior history of heart transplantation are not exclusion criteria if the inclusion criteria are otherwise met.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with 1) advanced heart failure and 2) who have been admitted to the hospital, will be recruited from inpatient cardiology floors.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage change in skeletal muscle thickness from admission to nadir of muscle thickness | Images obtained at baseline after consent; then days 3 and 7 after baseline study visit; then every 7 days thereafter until end of the index hospitalization (until discharge or death)
  Quantify the percentage change in skeletal muscle thickness from admission to nadir of muscle thickness and describe the time course of muscle loss. We hypothesize that all patients will experience a decrease in skeletal muscle thickness in the days-to-weeks after admission, as indicated by change in skeletal muscle thickness on ultrasound, and anticipate the magnitude of this muscle thickness change to be in the range of -5%. This aim will be investigated in both patients who ultimately receive the HT or LVAD advanced therapies, and also those who do not.
Percentage change in skeletal muscle thickness after advanced therapies | Images obtained at baseline after consent; then days 3 and 7 after baseline study visit; then every 7 days thereafter until end of the index hospitalization (until discharge or death)
  Quantify the percentage change in skeletal muscle thickness achieved early after advanced therapies (LVAD/HT). We hypothesize that hospitalized patients with advanced heart failure will experience a minor muscle recovery during the hospital stay following advanced therapy surgeries, but not a recovery in the range of +5% which would likely require a 3-month follow-up period.
Relationship between muscle mass loss during cardiogenic shock and subsequent clinical outcomes | Images obtained at baseline after consent; then days 3 and 7 after baseline study visit; then every 7 days thereafter until end of the index hospitalization (discharge or death)
  Evaluate the relationship between muscle mass loss during cardiogenic shock and subsequent clinical outcomes. We hypothesize that a greater negative percent change in muscle thickness from admission to the nadir thickness value will be associated with higher inhospital mortality, and for those who receive an LVAD/HT a longer post-operative length of stay and greater probably of discharge to a rehabilitation facility as opposed to home.

SECONDARY OUTCOMES:
Geriatric nutritional risk index (GNRI) | Once at baseline
  Evaluating the association between malnutrition risk as assessed by geriatric nutritional risk index (GNRI) on admission and change in skeletal muscle thickness from admission to nadir.
Upper extremity versus lower extremity US muscle thickness decreases | Images obtained at baseline after consent; then days 3 and 7 after baseline study visit; then every 7 days thereafter until end of the index hospitalization (discharge or death)
  Determine if an upper extremity or lower extremity US muscle site location for percentage change is most strongly associated with mortality and with GNRI on admission.
Inhospital mortality | Index Hospitalization
  Occurence of mortality during index hospitalization
Post-LVAD/HT length of stay | Index Hospitalization
  Days from LVAD/HT surgery until discharge from hospital or death
Discharge to a rehabilitation facility versus home | Conclusion of index Hospitalization
  Discharge destination at conclusion of index hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No